CLINICAL TRIAL: NCT04919759
Title: Development, Implementation and Evaluation of Technology Mediated Lifestyle Intervention for Promoting Weight Loss and Improving Nutrition Behaviors Among Young Adults
Brief Title: Feasibility of Technology Mediated Lifestyle Intervention for Overweight and Obese Young Adults
Acronym: Rashakaty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Arab Emirates University (Other)
Collaborators: University of Sharjah (Other)
Responsible Party: Principal Investigator, Habiba I. Ali, Associate Professor, United Arab Emirates University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33/2014/2015
Record Dates: First submitted 2021-05-30; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Basic Blue K

STUDY DESIGN:
Intervention Model Description: Two arms, non-randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rashakaty Basic (R-Basic) (Active Comparator): Participants in the R-Basic intervention arm had access to a website that contained the study questionnaires and nutrition education materials
  Interventions: Behavioral: R-Basic
- Rashakaty Enhanced (R-Enhanced) (Experimental): Participants in the R-Enhanced intervention were given access to smart phones applications for monitoring diet and physical activity levels as well as an online access to a nutritionist
  Interventions: Behavioral: R-Enhanced

INTERVENTIONS:
Behavioral: R-Basic — Participants in the R-Basic arm received access to a static website that contained educational materials on healthier eating and physical activity and the study questionnaires. The R-Basic intervention was implemented in the University of Sharjah.
  Other Names: Rashakaty Basic intervention
  Arms: Rashakaty Basic (R-Basic)
Behavioral: R-Enhanced — The R-Enhanced intervention was guided by the Social Cognitive Theory and employed a variety of behavior modification strategies, including self-monitoring, goal setting, self-efficacy, and social support to facilitate changes in diet and physical activity. In addition, participants in the R-Enhanced intervention had online access to a nutritionist. The R-Enhanced intervention was implemented in the United Arab Emirates University.
  Other Names: Rashakaty Enhanced intervention
  Arms: Rashakaty Enhanced (R-Enhanced)

SUMMARY:
Rashakaty (Fitness for Me) study aimed to design a new technologies-based intervention using a website and smart phone applications and to test the feasibility of implementing a lifestyle intervention using these technologies for overweight and obese university students. The intervention was implemented in two universities in the United Arab Emirates

DETAILED DESCRIPTION:
Poor eating habits and sedentary lifestyle are common among young adults and increase risk for chronic diseases in subsequent years of life. Rashakaty (Fitness for Me) study aimed to design a new technologies-based intervention using a website and smart phone applications and to test the feasibility of implementing a lifestyle intervention using these technologies for overweight and obese university students. The study intervention was guided by Social Cognitive Theory. The study involved the development of a website, integrating educational material and mobile applications for monitoring diet and physical activity and a16-week feasibility trial to promote weight loss, improve food choices and increase physical activity levels. The trial consisted of two arms: Rashakaty Basic (R-Basic) and Rashakaty Enhanced (R-Enhanced).

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese (BMI ≥25.0
* Adults: Female
* Age: 18-35 years
* Current user of a smart phone
* Student in one of the two target universities in the United Arab Emirates
* Living in or off the university campus

Exclusion Criteria:

* Past or planned weight loss surgery
* Pregnant or breastfeeding
* Lost 7 kg in the past 3 months
* Following any weight loss program for 3 months or more
* Taking any steroid or thyroid hormones treatment or any other medication that may affect body weight
* Enrolled in medical and nutrition programs since one of the program components was nutrition knowledge assessments

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 246 (Actual)
Dates: Start 2016-08-21 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Body weight | 16 weeks
  changes in body weight
Body composition | 16 weeks
  Changes in body composition (percent body fat)

SECONDARY OUTCOMES:
Nutrition knowledge | 16 weeks
  The General Nutrition Awareness Questionnaire (GNKQ) validated by Parmenter and Wardle in the UK. was used after local adaptation. Four main categories containing a total of 58 items were assessed:1) Awareness of dietary recommendations (11 items); 2) Knowledge of sources of nutrients (37 items); (3) Using the information to make dietary choices (5 items); and 4) Awareness of diet-disease relationships (5 items).
Physical activity | 16 weeks
  Changes in physical activity (number of days and duration) was used using The International Physical Activity Questionnaire (IPAQ) - Short Form
Perceived social support from family and closest friends. | 16 weeks
  Perceived social support for healthier foods and physical activity scale of Health Beliefs Questionnaire which was originally developed by Anderson, E. and colleagues was used after adaptation for university students in the UAE. The social support subscale (16 items for healthy eating and 7 items for physical activity) measures social influences on participants by their family members and closest friends. Each question is scored 1-5 (1 - Strongly disagree, 5 - Strongly agree).
Perceived self-efficacy for healthier eating and physical activity | 16 weeks
  Perceived self-efficacy scale of Health Beliefs Questionnaire which was originally developed by Anderson, E. and colleagues after local adaptation was used. It consists of 33 items for healthy eating and 24 items for physical activity. The healthy food efficacy measure assesses the respondent's confidence in reducing fat, reducing sugar consumption and increasing fruit and vegetable intake. The physical activity measure consists of two subscales: overcoming barriers to engaging in physical activity and integrating physical activity into the daily routine. Each question is scored 0 to 100 (certain I cannot) to 100) all or most of the time.

CONTACTS AND LOCATIONS:
Overall Officials: Habiba I Ali, PhD, RD, CDE, Principal Investigator — United Arab Emirates University
Locations (1):
- United Arab Emirates University, Al Ain City, Select State Or Region, United Arab Emirates